CLINICAL TRIAL: NCT05337059
Title: Feasabilty and Physiological Effects of a Ventilation Strategy Combining PEEP and Tidal Volume Titration According to Inspiratory and Expiratory Transpulmonary Pressures in ARDS Patients..
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A03242-55
Record Dates: First submitted 2022-03-29; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: ARDS, Human
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Intervention Model Description: feasibility, monocentric, prospective study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transpulmonary based ventilation strategy (Experimental): PEEP and tidal volume will be set to target expiratory and inspiratory transpulmonary pressures of 0 and 20 cmH2O, respectively.
  Interventions: Other: PEEP and Tidal Volume Titration

INTERVENTIONS:
Other: PEEP and Tidal Volume Titration — PEEP and Tidal Volume Titration According to Inspiratory and Expiratory Transpulmonary Pressures

SUMMARY:
Expiratory or inspiratory transpulmonary pressures have been proposed to optimize ventilator settings in patients with ARDS. The aim of this study is to assess the feasibility and the physiological effects of a new method based on both expiratory and inspiratory transpulmonary pressures.

DETAILED DESCRIPTION:
Expiratory or inspiratory transpulmonary pressures have been proposed to optimize ventilator settings in patients with ARDS. A positive expiratory transpulmonary pressure may be considered as a target to limt the risk of collapse in dependant lung regions. Some authors propose to titrate PEEP to target an inspiratory transpulmonary pressure of 20cmH20 to limit the risk of overdistension in non-dependant regions.The aim of this study is to assess the feasibility and the physiological effects of a new method based on both expiratory and inspiratory transpulmonary pressures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Moderate to severe ARDS
* Written informed consent obtained from patient' surrogates

Exclusion Criteria:

* Pneumothorax
* Known pregnancy
* Contraindication to electrical impedance tomography or esophageal pressure measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Ventilation strategy failure | 48 hours
  Number of patients with failure criteria (barotrauma, hemodynamic failure, rescue therapy or acidemia)

SECONDARY OUTCOMES:
Short term physiologicals effects on hemodynamics | 45 minutes
  Cardiac index assed by Echocardiography (L/min/m^2)
All-cause mortality at day 28 | 28 days
  All-cause mortality
Ventilator-free days at day 28 | 28 days
  Number of alive ventilator free days
Short term physiologicals effects on respiratory mechanics | 45 minutes
  recruited lung volume (mL)
Short term physiologicals effects on gas exchange | 45 minutes
  PaO2/FiO2 ratio (mmHg)
Short term physiologicals effects on gas exchange | 45 minutes
  VD/VT
Short term physiologicals effects on gas exchange | 45 minutes
  PaCO2 (mmHg)
Short term physiologicals effects on respiratory mechanics | 45 minutes
  distribution of ventilation assed by electrical impedance tomography (COV, %)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No